CLINICAL TRIAL: NCT05953233
Title: School Inner City Air Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Boston Children's Hospital (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Peggy S Lai, Associate Professor, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: IRB-P00045373; R21AI178155 (NIH)
Record Dates: First submitted 2023-06-27; First posted 2023-07-20 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Viral Infection
MeSH Terms: conditions — Virus Diseases

STUDY DESIGN:
Intervention Model Description: Classrooms will be randomized in a 1:1 ratio using a random number generator to active vs sham HEPA arms
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Sham cleaners are constructed by removing the filters from air cleaners and adding a sound generator rendering them indistinguishable from active HEPA cleaners.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active HEPA cleaner (Experimental): Active HEPA cleaners will be placed in classrooms throughout the school year
  Interventions: Other: Active classroom HEPA cleaner
- Sham HEPA cleaner (Placebo Comparator): Sham HEPA cleaners will be placed in classrooms throughout the school year
  Interventions: Other: Sham classroom HEPA cleaner

INTERVENTIONS:
Other: Active classroom HEPA cleaner — Commercially available portable HEPA cleaner
  Arms: Active HEPA cleaner
Other: Sham classroom HEPA cleaner — Commercially available portable HEPA cleaner with filtration device removed
  Arms: Sham HEPA cleaner

SUMMARY:
The goal of this randomized clinical trial is to test the efficacy of high efficiency particulate air (HEPA) cleaners in reducing respiratory viral exposure and infections in elementary school classrooms. Classrooms will be randomized to active vs. sham HEPA cleaners. The main questions it aims to answer are:

* Do classroom HEPA cleaners reduce exposure to viruses?
* Do classroom HEPA cleaners reduce student and teacher infections?
* Do classroom HEPA cleaners reduce infections in family members?

DETAILED DESCRIPTION:
Classrooms from participating schools will be randomized to active vs. sham HEPA cleaners. From enrolled classrooms, we will enroll students, teachers, and members of the household. We will collect the following:

* longitudinal classroom air samples
* longitudinal upper respiratory samples
* longitudinal symptom surveys using the Wisconsin Upper Respiratory Symptom Survey (WURSS) Viral testing on collected air and respiratory samples will be performed using digital polymerase chain reaction (dPCR).

ELIGIBILITY:
Inclusion Criteria:

Children

* Grades K-5 (age 6-12 years)
* Attend one of the schools that the study team has permission to obtain classroom/school environmental samples
* Have no plans to move schools within the upcoming 12 months
* Subject and/or parent guardian must be able to understand and provide informed consent and also willing to participate in the study

Adults

* Adult (age 21 or older) parent, caretaker, or household member of child participating in this study, or teacher in classroom participating in study
* Able to understand and provide informed consent

Exclusion Criteria:

Children

* Contraindication to or inability to participate in home self-collection of nasal swab samples
* Severe chronic diseases (e.g. cancer, genetic or congenital disorders interfering with mobility)
* Severe neurobehavioral, neurodevelopmental or psychiatric disorders requiring special assistance
* Families who do not speak English or Spanish well enough to complete the survey questions, as validated versions in other languages are not available for all of the measures

Adults

* Contraindication to or inability to participate in home self-collection of nasal swab samples
* Severe chronic diseases (e.g. cancer, genetic or congenital disorders interfering with mobility)
* Severe neurobehavioral, neurodevelopmental or psychiatric disorders requiring special assistance
* Families who do not speak English or Spanish well enough to complete the survey questions, as validated versions in other languages are not available for all of the measures

Ages: 6 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-09-15 (Actual); Primary Completion 2029-08 (Estimated); Study Completion 2030-08 (Estimated)

PRIMARY OUTCOMES:
Viral pathogen detected in upper respiratory sample | 1 year
  Presence/absence of a respiratory virus in upper respiratory sample

SECONDARY OUTCOMES:
Symptomatic respiratory infection (student, teacher) | 1 year
  Presence/absence of a cold based on 30 day recall
Symptomatic respiratory infection (household member) | 1 year
  Presence/absence of a cold based on 30 day recall
Viral detection in classroom bioaerosol sample | 1 year
  Viral detection in classroom bioaerosol sample (viral copy number per cubic meter of air)
Severity of a cold in child using the WURSS-K - Kids Daily Symptom Report | 1 year
  Severity of a cold (when present) in child will be graded using the Wisconsin Upper Respiratory Symptom Survey Kids Daily Symptom Report (WURSS-K). Range 0 - 42; higher indicates more severe.
Severity of a cold in adult using the WURSS-24 | 1 year
  Severity of a cold (when present) in adult will be graded using the Wisconsin Upper Respiratory Symptom Survey 24 Daily Symptom Report (WURSS-24). Range 0 - 161; higher indicates more severe.
Number of missed school or work days in last 30 days | 1 year
  30 day recall of missed school or work days. Range 0 - 30; higher indicates more severe.
Number of days requiring inpatient or outpatient care in last 30 days | 1 year
  30 day recall of healthcare utilization defined as number of days requiring outpatient or inpatient hospital care. Range 0 - 30; higher indicates more severe.

CONTACTS AND LOCATIONS:
Locations (1):
- Mass General Brigham, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided
The data will be made openly available through BioLINCC consistent with privacy and informed consent. As above, released individual-level data will not include information that alone or in conjunction with other data could readily identify individual participants. These data will be summarized and aggregated before sharing in BioLINCC. Data from research participants who refused to permit data sharing will be removed from the repository data set. All study data will be preserved as per study consents.